CLINICAL TRIAL: NCT06893536
Title: Impact of Perioperative Nutritional Status and Management in the Context of Resectable Pancreatic Adenocarcinoma
Acronym: PAAD
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9062
Record Dates: First submitted 2024-07-04; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2024-07

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Pancreatic Adenocarcinoma; Digestive tract; Hypercatabolism; Malnutrition,
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with pancreatic adenocarcinoma are frequently in a situation of malnutrition, in a context of functional alteration of the digestive tract, and hypercatabolism.

As a result, nutritional support is frequently necessary perioperatively, but currently does not follow a specific protocol, and without coordination.

It then appears the need to evaluate the prevalence of malnutrition, its impact on perioperative morbidity and mortality, and current management methods.

Depending on the findings, subsequent interventional studies will be carried out on the subject, exploring the different modalities of artificial nutrition.

ELIGIBILITY:
Inclusion Criteria:

* Major subject (≥18 years old)
* Subject with pancreatic adenocarcinoma authenticated by pathology
* Subject candidate for curative surgical treatment
* Subject operated on in the visceral and digestive surgery department, NHC Strasbourg, during the period from January 1, 2018 to December 31, 2022
* Absence of written opposition in the subject's medical file to the reuse of their data for scientific research purposes.

Exclusion criteria:

* Subject having expressed opposition to participating in the study
* Subject presenting a metastatic form or one not accessible to surgical treatment considered curative of pancreatic adenocarcinoma
* Subject under guardianship or curatorship
* Subje

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major subject (≥18 years old) with pancreatic adenocarcinoma authenticated by pathology and operated on in the visceral and digestive surgery department, NHC Strasbourg, during the period from January 1, 2018 to December 31, 2022
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10-12 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10-12 (Estimated)

PRIMARY OUTCOMES:
Study of the Severity of Perioperative Malnutrition in Pancreatic Adenocarcinoma | Up to 1 year
  The CCI score measures a patient's postoperative outcome based on the number and severity of complications occurring on a scale of 0 to 100:
  0: No complications 100: Death

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Chirurgie Viscérale et Digestive - CHU de Strasbourg - France, Strasbourg, France